CLINICAL TRIAL: NCT00273455
Title: Lumigan Versus Cosopt
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pharmaceutical Research Network (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PRN 05-017
Record Dates: First submitted 2006-01-06; First posted 2006-01-09 (Estimated); Last update posted 2008-11-19 (Estimated); Status verified 2008-11

CONDITIONS: Open-Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — dorzolamide; Timolol

INTERVENTIONS:
Drug: bimatoprost 0.03%
Drug: dorzolamide 2%/timolol maleate 0.5% fixed combination
Drug: placebo

SUMMARY:
To compare the intraocular pressure effect and safety of the dorzolamide/timolol fixed combination given twice daily versus bimatoprost given once every evening in patients with open-angle glaucoma in patients insufficiently controlled on latanoprost monotherapy

ELIGIBILITY:
Inclusion Criteria:

* adults with a diagnosis of bilateral open-angle glaucoma including: primary, pigment dispersion or exfoliation in both eyes
* on no therapy the intraocular pressure should be 22-29 mm Hg inclusive at the 8:00 AM measurement
* visual acuity should be 20/200 or better in each eye

Exclusion Criteria:

* historical failure to respond to topical beta-blockers in a clinically meaningful manner
* any contraindication to study medications
* any anticipated change, or modification in the 6 weeks prior to Visit 1, in systemic hypertensive therapy during the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34
Dates: Start 2006-01; Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William C. Stewart, MD, Study Director — Pharmaceutical Research Network, LLC; Robert D. Williams, MD, Principal Investigator — Taustine Eye Center; Robert H. Stewart, MD, Principal Investigator — Houston Eye Associates; Elizabeth D. Sharpe, MD, Principal Investigator — Glaucoma Consultants & Center for Eye Research, PA
Locations (3):
- United States (3):
  - Taustine Eye Center, Louisville, Kentucky
  - Glaucoma Consultants & Center for Eye Research, PA, Mt. Pleasant, South Carolina
  - Houston Eye Associates, Houston, Texas